CLINICAL TRIAL: NCT04875858
Title: Non-randomized Clinical Trial to Compare the Immunogenicity of Revaccination With 23-valent Pneumococcal Polysaccharide Vaccine Between Healthy Elderly and Those With Diabetes in Korea
Brief Title: Immunogenicity After Revaccination With 23-valent Pneumococcal Polysaccharide Vaccine: Healthy Elderly People Versus Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joon Young Song, Professor, Korea University Guro Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020GR0143
Record Dates: First submitted 2020-11-24; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pneumococcal Infections
Keywords: Streptococcus pneumoniae; Diabetes Mellitus; Immunogenicity, Vaccine; Pneumococcal Vaccines
MeSH Terms: conditions — Pneumococcal Infections; Diabetes Mellitus | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy old adults aged 70-75 years who received PPSV23 (Active Comparator): Recruitment of 254 healthy 70-75-year healthy old adults who meet the selection and exclusion criteria and voluntarily agree to participate in this study. Vaccination -Based on guidelines for vaccination. Injecting muscles on the triceps Visit 4 weeks after vaccination ․ Blood sample collection for evaluation of immunogenicity (10 mL) ․ Comparison of GMT and seroconversion rates of IgG antibody titers against 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F and 23F) -Comparison of GMT and seroconversion rates of opsonophagocytic killing assay (OPA) for four pneumococcal serotypes (serotypes 5, 6B, 18C, 19A)
  Interventions: Drug: ProDiax-23 (PPSV23)
- old adults who have diabetes mellitus aged 70-75 years who rec (Experimental): Recruitment of 254 healthy 70-75-year diabetic old adults who meet the selection and exclusion criteria and voluntarily agree to participate in this study. Vaccination -Based on guidelines for vaccination. Injecting muscles on the triceps Visit 4 weeks after vaccination ․ Blood sample collection for evaluation of immunogenicity (10 mL) ․ Comparison of GMT and seroconversion rates of IgG antibody titers against 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F and 23F) -Comparison of GMT and seroconversion rates of opsonophagocytic killing assay (OPA) for four pneumococcal serotypes (serotypes 5, 6B, 18C, 19A)
  Interventions: Drug: ProDiax-23 (PPSV23)

INTERVENTIONS:
Drug: ProDiax-23 (PPSV23) — diabetic old adults aged 70-75 years who received PPSV23 in previous 5-7 years (Persons 65-70 years old who have been inoculated with PPSV23 and 5-7 years have passed) and healthy old adults aged 70-75 years who received PPSV23 in previous 5-7 years (Persons 65-70 years old who have been inoculated with PPSV23 and 5-7 years have passed)

SUMMARY:
Pneumococcal disease causes thousands of infections, such as meningitis, bloodstream infections, pneumonia, and ear infections in US annually. As pneumococcal vaccines provide serotype-specific protection, it is important to induce sufficient immune responses for the most clinically relevant serotypes. All adults aged 65 years or older are recommended to receive PPSV23 vaccination irrespective of underlying medical conditions. Thus, since May 2013, South Korea introduced PPSV23 in the national immunization program for elderly individuals aged ≥65 years. Following PPSV23 vaccination, serotype-specific IgG concentrations and OPA titers increase and then decline over time thereby decreasing protective efficacy, although these might remain above pre-vaccination levels until 5 years from PPSV23 administration. The decline of pneumococcal immunity may be more prominent among chronically ill patients, including those with diabetes. Currently however, revaccination is not recommended. In this study, we aimed to evaluate the serotype specific immunogenicity between healthy elderly people and old adults with diabetes after revaccination with PPSV23 at the age of 70-75 years. Serotype-specific IgG concentrations and opsonophagocytic killing activity (OPA) titers will be assessed.

ELIGIBILITY:
Inclusion Criteria

* Elderly people aged 70-75 years
* Had received PPSV23 in the previous 5-7 years

Exclusion Criteria:

* Immunocompromised patients
* Subjects receiving immunosuppressive agents
* Subjects with a history of vaccination with pneumococcal conjugate vaccine
* Subjects with a history of pneumococcal disease (positive culture from blood or other sterile fluid)
* Fever (defined as an oral temperature >37.5℃) within 24 h before PPSV23 vaccination

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Serotype-specific immunogenicity assessed by opsonophagocytic killing assay. | up to one month after vaccination
  After PPSV23 vaccination, blood samples (10 mL) will be collected before vaccination and at 4 weeks post-vaccination. Serotype-specific opsonophagocytic activity (OPA) will be evaluated from those blood samples by opsonophagocytic killing assay for 4 serotypes (5, 6B, 18C, 19A).

SECONDARY OUTCOMES:
Serotype-specific IgG antibody concentrations assessed by ELISA. | up to one month after vaccination
  After PPSV23 vaccination, blood samples (10 mL) will be collected before vaccination and at 4 weeks post-vaccination. Serotype-specific IgG antibody concentrations for 13 serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, 22F and 23F) will be measured.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to one month after vaccination
  Solicited local or systemic reactions to the vaccines will be monitored using diary cards during the14 days post-vaccination. Participants will be asked to record pain, tenderness and redness diameter at both injection sites and systemic symptoms such as headache, malaise, chills, muscle aches, and arthralgia. Severity will be recorded according to the Food and Drug Administration Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Subjects will be also asked to record any unsolicited adverse event during the 14 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Young Song, MD, PhD., Principal Investigator — Professor
Locations (1):
- Koera University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song JY, Cheong HJ, Tsai TF, Chang HA, Choi MJ, Jeon JH, Kang SH, Jeong EJ, Noh JY, Kim WJ. Immunogenicity and safety of concomitant MF59-adjuvanted influenza vaccine and 23-valent pneumococcal polysaccharide vaccine administration in older adults. Vaccine. 2015 Aug 26;33(36):4647-52. doi: 10.1016/j.vaccine.2015.05.003. Epub 2015 May 14. PMID 25980426
- [Background] Kawakami K, Kishino H, Kanazu S, Toshimizu N, Takahashi K, Sterling T, Wang M, Musey L. Revaccination with 23-valent pneumococcal polysaccharide vaccine in the Japanese elderly is well tolerated and elicits immune responses. Vaccine. 2016 Jul 19;34(33):3875-81. doi: 10.1016/j.vaccine.2016.05.052. Epub 2016 Jun 10. PMID 27265450
- [Background] Choi WS, Choi JH, Kwon KT, Seo K, Kim MA, Lee SO, Hong YJ, Lee JS, Song JY, Bang JH, Choi HJ, Choi YH, Lee DG, Cheong HJ; Committee of Adult Immunization; Korean Society of Infectious Diseases. Revised adult immunization guideline recommended by the korean society of infectious diseases, 2014. Infect Chemother. 2015 Mar;47(1):68-79. doi: 10.3947/ic.2015.47.1.68. Epub 2015 Mar 30. No abstract available. PMID 25844267